CLINICAL TRIAL: NCT06974877
Title: A Phase 1 Study of Repeat PET/CT Imaging in People With CAPS and Anakinra-Induced Amyloidosis Using Amyloid-Reactive Peptide 124I-AT-01 (124I-p5+14, Iodine-124I-Evuzamitide) to Measure Changes in Organ-Specific Amyloid Load
Brief Title: Repeat PET/CT Imaging in People With CAPS and Anakinra-Induced Amyloidosis Using an Amyloid-Reactive Peptide to Measure Changes in Organ-Specific Amyloid Load
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 10001867; 001867-I
Record Dates: First submitted 2025-05-15; First posted 2025-05-16 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-05-08

CONDITIONS: Cryopyrin-Associated Periodic Syndromes; Amyloidosis
Keywords: Muckle-Wells Syndrome; Neonatal Onset Multisystem Inflammatory Disease; Interleukin 1 Receptor Antagonist Protein; Anakinra; AMYLOIDOSIS; AIL1RAP
MeSH Terms: conditions — Cryopyrin-Associated Periodic Syndromes; Amyloidosis

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Interventional (Experimental): Participants aged 18 years and older with anakinra-type amyloidosis (n=10) will be recruited from NIH protocol 17-I-0016. Upon confirmation of eligibility, they will undergo a PET/CT scan with the investigational radiotracer 124I-AT-01, which selectively binds to amyloid fibers. Blood and urine will also be collected for clinical and research analyses, including measurement of IL-1RA and other biomarkers. These scans and sample collections will be repeated about once every 6 months for 2 years.
  Interventions: Drug: 124I AT-01

INTERVENTIONS:
Drug: 124I AT-01 — 124I-AT-01 is an amyloid-reactive synthetic 45-L amino acid polypeptide radiolabeled with iodine-124, with a theoretical molecular weight of 4763.6 Da (based on amino acid sequence). The polypeptide, AT-01, is not pharmacologically active. 124I-AT-01 binds many forms of human and murine amyloid and is intended to be a PET imaging agent for the detection of amyloid deposits.

SUMMARY:
Background:

Anakinra is a drug used to treat people with certain diseases that affect their immune systems. Sometimes anakinra can cause proteins under the skin to clump together. These clumps are called amyloidosis; they can spread to other organs. The only way to diagnose amyloidosis is to remove a piece of tissue (biopsy). Researchers want to find a way to locate amyloidosis in internal organs using positron emission tomography (PET)/computed tomography (CT).

Objective:

To test a new tracer used during PET/CT scans in people with amyloidosis. A tracer is a radioactive dye injected into the body.

Eligibility:

Adults aged 18 years or older with amyloidosis from anakinra injections. They must be enrolled in NIH protocol 17-I-0016.

Design:

Participants will come to the clinic once every 6 months for 2 years. Each visit will be 1 day.

They will have a PET/CT scan with the new tracer at each visit: The tracer will be given through a tube attached to a needle inserted into a vein.

The PET/CT scanner is a machine shaped like a doughnut. Participants will lie still on a padded table. The table will move in and out of the machine. The scan takes about 1 hour.

Radiation from the tracer will remain in the body for 24 hours after each scan. Participants will need to follow rules to avoid exposing pets and other people.

Participants will collect a 24-hour urine sample before each visit. They will also have blood tests and a physical exam at each visit.

Participants will receive a follow-up phone call about 1 week after each visit.

DETAILED DESCRIPTION:
Study Description:

This is a phase 1 study to evaluate the feasibility of an investigational positron emission tomography (PET)/computed tomography (CT) radiotracer, 124I-AT-01, to screen for anakinra-induced amyloidosis in people with the cryopyrin-associated autoinflammatory syndromes (CAPS) (Muckle-Wells syndrome [MWS] or neonatal onset multisystem inflammatory disease [NOMID]), and to follow resolution of amyloidosis. This radiotracer binds to amyloid, so a PET/CT scan can show the presence and relative magnitude of amyloid.

Participants aged 18 years and older who developed local skin or systemic amyloidosis as a result of anakinra treatment will be recruited. They will have a PET/CT scan with radiotracer 124I-AT-01 about once every 6 months for 2 years. Blood and urine will be collected for clinical safety analyses, but no specimen will be collected for research or storage purposes.

The 124I-AT-01 PET/CT imaging is expected to be able to detect anakinra-induced amyloid in the skin and other organs (such as kidney, liver, and spleen). The percent change in quantitative uptake of 124I-AT-01 from baseline to each subsequent scan is expected to correlate with changes in clinical features related to load of amyloid in the body.

Primary Objectives:

1. To screen participants with fixed skin thickening at the site of anakinra injection and/or biopsy-proven anakinra-induced amyloidosis of the skin for the presence of systemic amyloidosis, using 124I-AT-01 PET/CT imaging.
2. To measure changes in organ-specific uptake of 124I-AT-01 from baseline in participants with anakinra-induced amyloidosis (local or systemic) using PET/CT imaging.
3. To assess the safety profile of 124I-AT-01 in participants with CAPS.

Primary Endpoints:

Change in organ-specific 124I-AT-01 uptake from baseline PET/CT imaging to the follow-up PET/CT imaging every 6 months for 2 years. Frequency of CAPS disease flares after exposure to 124I-AT-01.

ELIGIBILITY:
* INCLUSION CRITERIA:

An individual must meet all the following criteria to be eligible for this study:

1. Aged 18 years and older.
2. Currently enrolled on NIH protocol 17-I-0016 with a documented diagnosis of MWS or NOMID.
3. Agree to allow data collected in this study to be shared with and stored on NIH protocol 17-I-0016 for that study s research analyses.
4. Developed skin thickening at the site of anakinra injection.
5. Participants who can become pregnant or who can impregnate their partner must agree to use 2 highly effective methods of contraception, at least 1 of which must be a barrier method, when engaging in sexual activities that can result in pregnancy, beginning 28 days prior to baseline until 90 days after the last PET/CT scan. Acceptable methods of contraception include the following:

   1. Barrier methods:

      * External or internal condom with spermicide.
      * Diaphragm or cervical cap with a spermicide.
   2. Non-barrier methods:

      * Hormonal contraception.
      * Intrauterine device.
      * Hysterectomy, oophorectomy, or tubal ligation in women
      * Vasectomy in men
   3. Other.

EXCLUSION CRITERIA:

1. Known hypersensitivity to 124I-AT-01, AT-01, or any of their excipients.
2. Known hypersensitivity to KI.
3. Pregnant or breastfeeding.
4. Currently receiving dialysis.
5. Currently taking heparin or heparin derivatives (eg, low molecular weight heparins) or other blood thinners for anticoagulation.
6. Any condition that, in the opinion of the study team, contraindicates participation in this study.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-09-10 (Actual); Primary Completion 2031-07-01 (Estimated); Study Completion 2032-01-31 (Estimated)

PRIMARY OUTCOMES:
Change in organ-specific 124I AT-01 uptake from baseline PET/CT imaging to the follow up PET/CT imaging every 6 months for 2 years. | 2 years
  The gold standard for detecting amyloid deposits is tissue biopsy. With this compound, we expect to detect evidence of tissue deposits in the tissue at a much earlier stage and in a non invasive manner. By lowering the exposure to anakinra in participants with anakinra-associated systemic amyloidosis, the burden of amyloidosis is expected to reduce over time.
Frequency of CAPS disease flares after exposure to 124I AT 01. | Through end of study.
  This compound has not been used in patients with CAPS. We will monitor the participants to detect possible inflammatory disease flare following the exposure.

CONTACTS AND LOCATIONS:
Overall Officials: Sara Alehashemi, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
IPD will be shared in accordance with the NIH Data Management and Sharing Policy.
Time Frame: At the time of publication.
Access Criteria: Data will be shared in closed access repositories. PI will assess qualifications of other requests for data access.

REFERENCES:
- [Background] Alehashemi S, Dasari S, Metpally A, Uss K, Castelo-Soccio LA, Heller T, Kellman P, Chen MY, Ahlman M, Kim J, Wargo S, Kuhns DB, Fink D, de Jesus A, Martin PS, Chang R, Bolanos J, Lee CR, Nasr SH, Goldbach-Mansky R, McPhail E. Anakinra-Associated Systemic Amyloidosis. Arthritis Rheumatol. 2024 Jan;76(1):100-106. doi: 10.1002/art.42664. Epub 2023 Nov 29. PMID 37488949
- [Background] Nasr SH, Alehashemi S, Dasari S, Waldman M, Afzali B, Chiu A, Bolanos J, Goldbach-Mansky R, McPhail ED. Anakinra-associated renal amyloidosis. Kidney Int. 2024 Feb;105(2):395-396. doi: 10.1016/j.kint.2023.08.020. No abstract available. PMID 38245224
- [Background] Alehashemi S, Dasari S, de Jesus AA, Cowen EW, Lee CR, Goldbach-Mansky R, McPhail ED. Anakinra-Associated Amyloidosis. JAMA Dermatol. 2022 Dec 1;158(12):1454-1457. doi: 10.1001/jamadermatol.2022.2124. PMID 36223107
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_001867-I.html